CLINICAL TRIAL: NCT02540603
Title: Evaluation of a Full Face Mask for the Treatment of Obstructive Sleep Apnea (OSA) in NZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-179
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full Face Mask (Experimental): F&P Jupiter Full Face Mask with Headgear
  Interventions: Device: F&P Jupiter Full Face Mask

INTERVENTIONS:
Device: F&P Jupiter Full Face Mask — Investigative F&P Jupiter full face mask to be used for OSA therapy
  Other Names: Jupiter Mask

SUMMARY:
This investigation is designed to evaluate the performance (leak and comfort) as well as participant's overall acceptance of the investigative full face mask amongst OSA participants.

DETAILED DESCRIPTION:
A total number of up to 15 OSA participants who currently use full face masks will be recruited for the trial. Participants will be on the trial for three weeks, using the prototypes at home for two weeks. PAP baseline data on the participant's prescribed treatment pressure with their usual mask and will be collected for one week prior to mask fitting with the full face trial mask.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Diagnosed with OSA by a practicing physician
* Prescribed PAP therapy (Bi-Level or Continuous Positive Airway Pressure (CPAP) or Automatic Positive Airway Pressure (APAP))
* Existing full face users

Exclusion Criteria:

* Inability to give informed consent
* Patients who are in a coma or decreased level of consciousness
* Anatomical or physiological conditions making PAP therapy inappropriate (e.g unconsolidated facial fracture)
* Commercial Drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of CO2 retention
* Pregnant or think they may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with average system leak >60L/min | Two weeks in-home use
  Average system leak will be recorded through downloading of the data from the PAP device in L/min.

SECONDARY OUTCOMES:
Insights into mask fitting and removal. | Two weeks use
  Observations of the action of fitting the mask and removing the mask will be noted.
Number of participants that found the mask comfortable. | Two weeks in-home use
  Subjective feedback on comfort will be measured through questionnaires.

IPD SHARING:
Plan to Share IPD: No
Data will be shared to any other parties.